CLINICAL TRIAL: NCT04677296
Title: Clinical Trial to Compare the Efficacy and Safety of a Multiple Amino-acid Based ORS "VS002A" With the Standard WHO-ORS in the Management of Non-cholera Acute Watery Diarrhea in Infants and Young Children
Brief Title: Efficacy and Safety of "VS002A" With the Standard WHO-ORS in Non-cholera Acute Watery Diarrhea in Infants and Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Entrinsic Bioscience Inc. (Industry)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR-17028
Record Dates: First submitted 2020-11-17; First posted 2020-12-21 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Diarrhea, Infantile
MeSH Terms: conditions — Diarrhea, Infantile | interventions — World Health Organization oral rehydration solution

STUDY DESIGN:
Intervention Model Description: Randomized double blinded
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VS002A (Experimental): Amino acid based ORS/medical food (VS002A). Initial treatment dosing with VS002A will be estimated using body weight in accordance with 5-10 ml/kg after each loose stool as per icddr,b guidelines, to maintain ongoing loss.
  Interventions: Other: VS002A
- Standard WHO-ORS (Active Comparator): Standard WHO-ORS. Initial treatment dosing with WHO-ORS will be estimated using body weight in accordance with 5-10 ml/kg after each loose stool as per icddr,b guidelines, to maintain ongoing loss.
  Interventions: Other: WHO-ORS

INTERVENTIONS:
Other: VS002A — Amino acid based ORS/Medical food
  Arms: VS002A
Other: WHO-ORS — WHO Oral rehydration solution, which is glucose based
  Arms: Standard WHO-ORS

SUMMARY:
Randomized double blinded clinical trial comparing amino acid based oral rehydration solution/medical food and glucose-based oral rehydration solution is infectious diarrhea in pediatric population

ELIGIBILITY:
Inclusion criteria:

1. Age: 6 months - 36 months,
2. Duration of diarrhea ≤48 hours,
3. Some dehydration (judged clinically according to the "Dhaka method"),
4. Written informed consent by either parent/guardian.

Exclusion criteria:

1. Severe malnutrition (Weight-for-length WLZ/WHZ/WAZ <-3 or presence of nutritional edema)
2. Patients with diarrhea due to cholera.
3. Systemic illness (e.g. Pneumonia, tuberculosis, enteric fever, meningitis etc.)
4. Bloody diarrhea
5. Any congenital anomaly or disorder (e.g. diagnosed inborn error of metabolism, congenital cardiac disease, seizure disorders, hypothyroidism, Down's syndrome etc.)
6. Requirement of additional intravenous fluids after being provided with an IV for 4 hours on admission if severely dehydrated
7. Has documentation of taking antibiotic and/or antidiarrheal within the last 48 hours prior to hospitalization.

Ages: 6 Months to 36 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Measuring stool output on a diaper on female children will create a bias since it will be mixed with urine.
Enrollment: 312 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea in hospital (hours) | 5 days
  number of hours of diarrhea after randomization

SECONDARY OUTCOMES:
Stool output | 1 day
  Stool output in the 1st 24 hours of hospitalization (g/kg body wt.), divided into two 12-hour periods
Total stool output | 5 days
  Total amount of stool output during the study
ORS intake in the 1st 24 hours of hospitalization | 1 day
  Amount of intervention drink consumed in the first 24 hours after randomization
Total ORS intake | 5 days
  Amount of intervention drink consumed throughout the duration of the study
Unscheduled IV (frequency/ORS group) | 5 days
  Frequency of IV fluids between he 2 groups
Treatment failure (frequency/ORS group) | 5 days
  Frequency of treatment failures between the two groups
Output and frequency of vomiting | 5 days
  Amount and frequency of vomiting between the two groups
Change in body weight (between pre-randomization and post-treatment) | 5 days
  Body weight at randomization and post treatment
Urine output in the 1st 24 hours of hospitalization (g/kg body wt.) | 1 day
  Amount of urine in the first 24 hours after randomization
Total urine output during hospitalization | 5 days
  Total urine output (g/kg body wt.)
Documented infectious agent | 5 days
  Stool culture and recording of infectious agent causing the diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Tahmeed Ahmed, MD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Das R, Sobi RA, Sultana AA, Nahar B, Bardhan PK, Luke L, Fontaine O, Ahmed T. A double-blind clinical trial to compare the efficacy and safety of a multiple amino acid-based ORS with the standard WHO-ORS in the management of non-cholera acute watery diarrhea in infants and young children: "VS002A" trial protocol. Trials. 2022 Aug 25;23(1):706. doi: 10.1186/s13063-022-06601-5. PMID 36008819